CLINICAL TRIAL: NCT06899555
Title: REgistry of Paclitaxel Coated Drug Eluting Balloon in All Comers PaTients (REPEAT Registry)
Brief Title: REgistry of Paclitaxel Coated Drug Eluting Balloon in All Comers PaTients
Acronym: REPEAT
Status: Not yet recruiting | Type: Observational
Sponsor: Craigavon Area Hospital (Other)
Responsible Party: Principal Investigator, Dr I. B. A. Menown, Director, Interventional Research, Craigavon, Craigavon Area Hospital
Other Study IDs: TL/PMS/DEB/2024-01
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: CAD - Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Arm, 500 Patients

SUMMARY:
A post marketing, observational , multi centre, prospective registry to assess safety and performance of the Drug Eluting Balloon in patients undergoing percutaneous coronary intervention.

Rational : Although DEBs are generally considered safe, there remain many unanswered questions about DEB technology in a real-world population and only limited trial data from geographically or clinically diverse patient subgroups. To address some of the clinical and translational gaps in knowledge we thus plan a clinical registry to assess safety and performance of a novel design of a drug eluting

A real-world, all-comers coronary artery disease (CAD) population undergoing percutaneous coronary intervention (PCI) and suitable for treatment with a Paclitaxel Coated Coronary Balloon Dilatation Catheter.

Study Population - 500 Patients

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is a minimally invasive procedure treated as first line of treatment for symptomatic coronary artery disease (CAD). In 1977, Gruentzig performed the first balloon percutaneous transluminal coronary angioplasty (PTCA) but this was associated with acute dissection or elastic recoil and later restenosis (re-narrowing). Bare metal stents (BMS) were developed which helped address acute dissection or recoil but only modestly decreased the risk of restenosis (which still occurred in around 25% of people within six months).

Drug eluting stents (DES), coated with polymers which released drugs such as sirolimus or paclitaxel were then developed to reduce restenosis. Second-generation DES incorporating new metal platforms (changing from stainless steel to thinner strut metal alloys such as cobalt-chromium or platinum-chromium), new more biocompatible polymers, and new drugs such as Zotarolimus, Everolimus and Novolimus were associated with reduction in myocardial infarction (MI), target lesion revascularisation (TLR) and stent thombosis compared with first-generation DES.

However, even with second-generation DES, concerns remain regarding the risk of delayed healing, late stent thrombosis and in-stent restenosis (around 2% per year) and alteration of vascular physiology due to permanent caging by the stent. Hence, drug-eluting balloons (DEB), {also referred as Drug Coated Balloons (DCB)} were developed as a non-stent approach to circumvent some drawbacks of DES. Provided pre-dilatation does not induce excessive dissection or recoil requiring a stent, DEBs deliver rapid release and deposition of anti-restenotic drug in the vessel wall at the time of balloon inflation but without a permanent implant, thus enabling more rapid healing of the vessel, similar reduction in restenosis to DES but potentially reduced late complications.

Currently, DEBs are used in treating In-stent restenosis (ISR), bifurcation lesions, Ostial lesions, long & large lesions, De novo of small vessel disease, complex coronary interventions, and high bleeding risk situations. Although DEBs are generally safe and non-inferior to other contemporary treatment procedure there are many unanswered questions about DEB technology in real world population. Geographical distribution of clinical trials or sample size and diversification is an important criterion to evaluate the safety and efficacy of the DEBs in real- world settings. The trend indicates fewer domestic trials for DEB. In lieu of the above clinical and translational gaps a registry is planned to assess safety and performance of the Drug Eluting Balloon in CAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with symptomatic coronary artery disease (including those with acute coronary syndromes or Chronic Coronary Syndromes) with either symptoms and/or ischaemia.
* The patient must be able to understand and provide informed consent and comply with all study procedures.

Coronary angiographic inclusion criteria:

* ≥70% target lesion stenosis in LAD, LCX or RCA (or branches) which after successful pre-dilatation* has a residual stenosis ≤ 30% and no dissection of Type C or greater than (NHLBI guidelines)

  *pre-dilation permitted with SC or NC balloon catheter, cutting/scoring balloon, rotational/orbital atherectomy, or laser
* Target vessel reference diameter between 2.0 and 4.5 mm.

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) ≤ 30%
* Acute ST elevation MI (STEMI)
* Cardiogenic shock within 2 days prior to the index PCI.
* Known contraindication or hypersensitivity to paclitaxel, and/or to any anti-thrombotic and anti-platelet class of drugs
* Allergy to imaging contrast media which cannot be adequately pre-medicated.
* Patient undergoing planned surgery within 3 months with the necessity to stop dual antiplatelet therapy (DAPT).
* Patient is pregnant or breast feeding.
* Patient has received a heart transplant.
* Patient is unwilling or unable to give follow-up until study completion.
* Patient is currently participating in another trial.
* Life expectancy <1 year.

Angiographic exclusion criteria:

* Target lesion in the left main coronary artery.
* Flow limiting target vessel thrombus
* Vessel dissection requiring bailout stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A real-world, all-comers coronary artery disease (CAD) population undergoing percutaneous coronary intervention (PCI) and suitable for treatment with a Paclitaxel Coated Coronary Balloon Dilatation Catheter.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Target Lesion failure | 12 Month
  Target Lesion failure through 12-months [composite of cardiac death, target vessel myocardial infarction (MI) and ischaemia-driven target lesion revascularization (TLR)]

SECONDARY OUTCOMES:
Major Adverse Cardiac Event (MACE) | MACE at 1 year; Procedural & Device Success at Baseline
  Major Adverse Cardiac Event (MACE) [Time Frame: through 12 Months] - Composite of all cause death, any MI, any revascularization
  Device success [Time Frame: During index procedure] - Defined as the ability of the study device to be delivered, dilated and retrieved from the target lesion.
  Procedural success [Time Frame: From Index procedure till discharge] - Defined as technical and angiographic success in the absence of Major Adverse Cardiac Events (MACE) during hospitalization.

IPD SHARING:
Plan to Share IPD: No